CLINICAL TRIAL: NCT01606917
Title: Interventions for Lifestyle Changes to Promote Weight Reduction, a Randomized Controlled Trial in Primary Health Care
Acronym: LÄTTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Stefan Jansson, MD PhD Student, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OrebroCC
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Overweight/Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive lifestyle counseling (Experimental): Both dietary advice and individualized advice on increased regular physical activity.
  Interventions: Other: Intensive lifestyle counseling
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Intensive lifestyle counseling — Both dietary advice and individualized advice on increased regular physical activity
  Arms: Intensive lifestyle counseling

SUMMARY:
The purpose of this study is to examine the effects of a weight reduction program in adults, seen in a primary care setting, with overweight/obesity perceived as a health problem or with diseases related to overweight/obesity and ambitions to achieve weight reduction as part of treatment.

DETAILED DESCRIPTION:
Patients seeking advice for overweight/obesity or illness related to overweight/obesity at eight primary health care centers in Sweden were randomized either to intervention or control care groups with both dietary advice and individualized advice on increased regular physical activity. Main outcome measures were reduction in body weight of 5 percent or more from study start.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 70 years of age who consulted or were in care for overweight/obesity with or without type 2 diabetes
* Hypertension, CVD
* Coronary heart disease (CHD)
* Dyslipidemia
* Gallstone or musculoskeletal disorders

Exclusion Criteria:

* Patients were not eligible if they were already taking part in another weight control program
* Understood the Swedish language poorly
* Were mentally ill or had an alcohol or drug addiction.
* Nor were they eligible if they had a physical disability preventing intensified physical activity or were pregnant at study start.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2004-10; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieved target weight at two years | 2 years

SECONDARY OUTCOMES:
Clinical or laboratory manifestations of their baseline illness (type 2 diabetes, hypertension, CHD, dyslipidemia) or death of any cause. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan P.O Jansson, MD PhD student, Principal Investigator — Family Medicine Research Centre, Örebro County Council, School of Health and Medical Sciences, Örebro University
Locations (1):
- Orebro County Council, Örebro, Sweden

REFERENCES:
- [Derived] Jansson SP, Engfeldt P, Magnuson A, Pt GL, Liljegren G. Interventions for lifestyle changes to promote weight reduction, a randomized controlled trial in primary health care. BMC Res Notes. 2013 May 27;6:213. doi: 10.1186/1756-0500-6-213. PMID 23711165
- See also: Medicine Research Centre — http://www.orebroll.se/sv/Forskning/Forskningsomraden/Allmanmedicin1/